CLINICAL TRIAL: NCT05592509
Title: Evaluation of the Antioxidant Effect of a Mixture of Ozonated Vegetable Oil and Vitamin Complex (Vitamin K2 and Vitamin B9) in Moderately Active Subjects With "Physical Activity Level" (LAF: 1.70-1.99): Pilot Study
Brief Title: Antioxidant Effect of Ozonated Vegetable Oil and Vitamins in Moderately Active Subjects
Acronym: ANTIOX001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S&R Farmaceutici spa (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ANTIOX001
Record Dates: First submitted 2022-09-27; First posted 2022-10-24 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2022-10

CONDITIONS: Oxidative Stress; Inflammation
Keywords: ozonated sunflower oil; antioxidant; inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: Twenty subjects will be divided into two groups of 10 subjects following randomization. The first group will take the dietary supplement (three capsules per day) for 60 days, while the second group will take a placebo (three capsules per day) for 60 days.
  During the treatment period (60 days), the two groups will undergo follow-ups at days 0, 15, 30 and 60 within which clinical and hematochemical examinations will be conducted as per Table 2. At the end of the 60 days, after the wash-out period (two weeks), as per the cross-over design the group previously taking the dietary supplement will be on placebo (three capsules per day) for 60 days, while the group previously taking placebo will take the dietary supplement (three capsules per day) for 60 days. Again, follow-ups will be at 0, 15, 30 and 60 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement (Active Comparator): This arm will take dietary supplement
  Interventions: Dietary Supplement: Ozonized vegetable oil with vitamines
- Placebo (Placebo Comparator): Placebo will take the placebo
  Interventions: Dietary Supplement: Ozonized vegetable oil with vitamines

INTERVENTIONS:
Dietary Supplement: Ozonized vegetable oil with vitamines — description: A single capsule is composed by ozonized vegetable oil (75 mg), vitamin K2 (20 mcg), vitamin B9 (130 mcg). The posology is three capsules/day.
  The time of administration is two months.

SUMMARY:
The purpose of this pilot study is to evaluate the antioxidant effect of a nutraceutical formulation based on vegetable oil and vitamin complex (vitamin K2 and vitamin B9) in subjects with the same level of physical activity (LAF 1.70-1.99, normally active or moderately active).

DETAILED DESCRIPTION:
Study design: The pilot study will enroll 20 subjects with physical activity level LAF 1.70-1.99 (normally active or moderately active).

The 20 subjects will be divided into two groups of 10 subjects following randomization. The first group will take the dietary supplement (three capsules per day) for 60 days, while the second group will take a placebo (three capsules per day) for 60 days.

During the treatment period (60 days), the two groups will undergo follow-ups at days 0, 15, 30 and 60 within which clinical and hematochemical examinations will be conducted. At the end of the 60 days, after the wash-out period (two weeks), as per the cross-over design the group previously taking the dietary supplement will be on placebo (three capsules per day) for 60 days, while the group previously taking placebo will take the dietary supplement (three capsules per day) for 60 days. Again, follow-ups will be at 0, 15, 30 and 60 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes;
* Aged between 18 and 60 years, naïve to taking antioxidant supplements;
* Absent of chronic diseases and current therapies;
* willing and able to understand and sign an informed consent;
* willing to follow a dietary pattern developed according to the LARN (Reference Intake Levels of Nutrients and Energy for the Italian Population) guidelines that establish reference intake levels for Average Energy Requirement (AR) and Macronutrients (Carbohydrates, Lipids and Protein) for the Italian adult population [LARN Tables*];
* Hematobiochemical examinations in normal range: blood count, lipid status, renal and liver function, inflammatory status (Tnfα, C-reactive protein, ESR), glycemic profile (Fasting blood glucose, HbA1C, insulinemia, Homa Index);
* BMI in the normal range (18-24.99);
* Physical activity level LAF 1.70-1.99 (normally active or moderately active)

Exclusion Criteria:

* Chronic diseases (chronic renal failure, chronic hepatocellular failure, autoimmune diseases, chronic inflammatory bowel disease, diabetes mellitus, end-stage neoplasms, symptomatic chronic ischemic heart disease)
* Severe hypertension;
* High-grade hypercholesterolemia;
* Age < 18 years;
* Poor compliance;
* Intake of dietary supplements containing antioxidants;
* Untreated hypothyroidism;
* Pregnant and lactating women;
* Underweight subjects (BMI ≤18.49);
* Overweight subjects (25≤ BMI ≤30);
* Subjects with obesity (BMI ≥30);
* Subjects with different levels of physical activity: very active (LAF 2.00-2.40) and sedentary (LAF 1.40-1.69).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Evaluation of hematic oxidative stress by quantifying ROS (CARR U) | baseline value before crossover
  Evaluation of the ability of the dietary supplement to modulate oxidative stress over time by quantifying reactive oxygen metabolites (ROS) using CARR U as units of measure comparing with the placebo-treated group at each follow-up
Evaluation of hematic oxidative stress by quantifying ROS (CARR U) | evaluation after 15 days of treatment before crossover
  Evaluation of the ability of the dietary supplement to modulate oxidative stress over time by quantifying reactive oxygen metabolites (ROS) using CARR U as units of measure comparing with the placebo-treated group at each follow-up
Evaluation of hematic oxidative stress by quantifying ROS (CARR U) | evaluation after 30 days of treatment before crossover
  Evaluation of the ability of the dietary supplement to modulate oxidative stress over time by quantifying reactive oxygen metabolites (ROS) using CARR U as units of measure comparing with the placebo-treated group at each follow-up
Evaluation of hematic oxidative stress by quantifying ROS (CARR U) | evaluation after 60 days of treatment before crossover
  Evaluation of the ability of the dietary supplement to modulate oxidative stress over time by quantifying reactive oxygen metabolites (ROS) using CARR U as units of measure comparing with the placebo-treated group at each follow-up
Evaluation of hematic oxidative stress by quantifying ROS (CARR U) | baseline after crossover
  Evaluation of the ability of the dietary supplement to modulate oxidative stress over time by quantifying reactive oxygen metabolites (ROS) using CARR U as units of measure comparing with the placebo-treated group at each follow-up
Evaluation of hematic oxidative stress by quantifying ROS (CARR U) | evaluation after 15 days of treatment after crossover
  Evaluation of the ability of the dietary supplement to modulate oxidative stress over time by quantifying reactive oxygen metabolites (ROS) using CARR U as units of measure comparing with the placebo-treated group at each follow-up
Evaluation of hematic oxidative stress by quantifying ROS (CARR U) | evaluation after 30 days of treatment after crossover
  Evaluation of the ability of the dietary supplement to modulate oxidative stress over time by quantifying reactive oxygen metabolites (ROS) using CARR U as units of measure comparing with the placebo-treated group at each follow-up
Evaluation of hematic oxidative stress by quantifying ROS (CARR U) | evaluation after 60 days of treatment after crossover
  Evaluation of the ability of the dietary supplement to modulate oxidative stress over time by quantifying reactive oxygen metabolites (ROS) using CARR U as units of measure comparing with the placebo-treated group at each follow-up
Evaluation of hematic oxidative stress by quantifying biological antioxidant potential (umol/l) | Baseline before crossover
  Evaluation of the ability of the dietary supplement to modulate oxidative stress over time by quantifying biological antioxidant potential using umol/l as units of measure comparing with the placebo-treated group at each follow-up
Evaluation of hematic oxidative stress by biological antioxidant potential (umol/l) | evaluation after 15 days of treatment before crossover
  Evaluation of the ability of the dietary supplement to modulate oxidative stress over time by quantifying biological antioxidant potential using umol/l as units of measure comparing with the placebo-treated group at each follow-up
Evaluation of hematic oxidative stress by quantifying biological antioxidant potential (umol/l) | evaluation after 30 days of treatment before crossover
  Evaluation of the ability of the dietary supplement to modulate oxidative stress over time by quantifying biological antioxidant potential using umol/l as units of measure comparing with the placebo-treated group at each follow-up
Evaluation of hematic oxidative stress by quantifying biological antioxidant potential (umol/l) | evaluation after 60 days of treatment before crossover
  Evaluation of the ability of the dietary supplement to modulate oxidative stress over time by quantifying biological antioxidant potential using umol/l as units of measure comparing with the placebo-treated group at each follow-up
Evaluation of hematic oxidative stress by quantifying biological antioxidant potential (umol/l) | baseline after crossover
  Evaluation of the ability of the dietary supplement to modulate oxidative stress over time by quantifying biological antioxidant potential using umol/l as units of measure comparing with the placebo-treated group at each follow-up
Evaluation of hematic oxidative stress by quantifying biological antioxidant potential (umol/l) | evaluation after 15 days of treatment after crossover
  Evaluation of the ability of the dietary supplement to modulate oxidative stress over time by quantifying biological antioxidant potential using umol/l as units of measure comparing with the placebo-treated group at each follow-up
Evaluation of hematic oxidative stress by quantifying biological antioxidant potential (umol/l) | evaluation after 30 days of treatment after crossover
  Evaluation of the ability of the dietary supplement to modulate oxidative stress over time by quantifying biological antioxidant potential using umol/l as units of measure comparing with the placebo-treated group at each follow-up
Evaluation of hematic oxidative stress by quantifying biological antioxidant potential (umol/l) | evaluation after 60 days of treatment after crossover
  Evaluation of the ability of the dietary supplement to modulate oxidative stress over time by quantifying biological antioxidant potential using umol/l as units of measure comparing with the placebo-treated group at each follow-up

SECONDARY OUTCOMES:
Assessment of hematic inflammatory parameters by quantifying C-Reactive Protein (CRP) | baseline value before crossover
  Evaluation of the modulation of inflammatory parameters by C-Reactive Protein (CRP) using mg/dl as unit of measure
Assessment of hematic inflammatory parameters by quantifying C-Reactive Protein (CRP) | evaluation after 60 days of treatment before crossover
  Evaluation of the modulation of inflammatory parameters by C-Reactive Protein (CRP) using mg/dl as unit of measure
Assessment of hematic inflammatory parameters by quantifying C-Reactive Protein (CRP) | baseline after crossover
  Evaluation of the modulation of inflammatory parameters by C-Reactive Protein (CRP) using mg/dl as unit of measure
Assessment of hematic inflammatory parameters by quantifying C-Reactive Protein (CRP) | evaluation after 60 days of treatment after crossover
  Evaluation of the modulation of inflammatory parameters by C-Reactive Protein (CRP) using mg/dl as unit of measure
Assessment of hematic inflammatory parameters by quantifying Erythrocyte Sedimentation Rate (ESR) | baseline value before crossover
  Evaluation of the modulation of inflammatory parameters by measuring Erythrocyte Sedimentation Rate (ESR) using mm/h as unit of measure
Assessment of hematic inflammatory parameters by quantifying Erythrocyte Sedimentation Rate (ESR) | evaluation after 60 days of treatment before the crossover
  Evaluation of the modulation of inflammatory parameters by measuring Erythrocyte Sedimentation Rate (ESR) using mm/h as unit of measure
Assessment of hematic inflammatory parameters by quantifying Erythrocyte Sedimentation Rate (ESR) | baseline after crossover
  Evaluation of the modulation of inflammatory parameters by measuring Erythrocyte Sedimentation Rate (ESR) using mm/h as unit of measure
Assessment of hematic inflammatory parameters by quantifying Erythrocyte Sedimentation Rate (ESR) | evaluation after 60 days of treatment after crossover
  Evaluation of the modulation of inflammatory parameters by measuring Erythrocyte Sedimentation Rate (ESR) using mm/h as unit of measure
Assessment of hematic inflammatory parameters by quantifying Tumor Necrosis Factor (Tnfα) | baseline value before crossover
  Evaluation of the modulation of inflammatory parameters by quantifying Tumor Necrosis Factor (Tnfα) using pg/mL as unit of measure
Assessment of hematic inflammatory parameters by quantifying Tumor Necrosis Factor (Tnfα) | evaluation after 60 days of treatment before crossover
  Evaluation of the modulation of inflammatory parameters by quantifying Tumor Necrosis Factor (Tnfα) using pg/mL as unit of measure
Assessment of hematic inflammatory parameters by quantifying Tumor Necrosis Factor (Tnfα) | baseline after crossover
  Evaluation of the modulation of inflammatory parameters by quantifying Tumor Necrosis Factor (Tnfα) using pg/mL as unit of measure
Assessment of hematic inflammatory parameters by quantifying Tumor Necrosis Factor (Tnfα) | evaluation after 60 days of treatment after crossover
  Evaluation of the modulation of inflammatory parameters by quantifying Tumor Necrosis Factor (Tnfα) using pg/mL as unit of measure
Assessment of hematic inflammatory parameters by quantifying Cortisol level | baseline value before crossover
  Evaluation of the modulation of inflammatory parameters by measuring Cortisol level using μg/dl as unit of measure
Assessment of hematic inflammatory parameters by quantifying Cortisol level | evaluation after 60 days of treatment before crossover
  Evaluation of the modulation of inflammatory parameters by measuring Cortisol level using μg/dl as unit of measure
Assessment of hematic inflammatory parameters by quantifying Cortisol level | baseline value after crossover
  Evaluation of the modulation of inflammatory parameters by measuring Cortisol level using μg/dl as unit of measure
Assessment of hematic inflammatory parameters by quantifying Cortisol level | evaluation after 60 days of treatment after crossover
  Evaluation of the modulation of inflammatory parameters by measuring Cortisol level using μg/dl as unit of measure

CONTACTS AND LOCATIONS:
Overall Officials: Emanuela Floridi, Doctor, Principal Investigator — Crabion srl
Locations (1):
- Crabion srl, Corciano, Perugia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simioni C, Zauli G, Martelli AM, Vitale M, Sacchetti G, Gonelli A, Neri LM. Oxidative stress: role of physical exercise and antioxidant nutraceuticals in adulthood and aging. Oncotarget. 2018 Mar 30;9(24):17181-17198. doi: 10.18632/oncotarget.24729. eCollection 2018 Mar 30. PMID 29682215
- [Background] Powers SK, Deminice R, Ozdemir M, Yoshihara T, Bomkamp MP, Hyatt H. Exercise-induced oxidative stress: Friend or foe? J Sport Health Sci. 2020 Sep;9(5):415-425. doi: 10.1016/j.jshs.2020.04.001. Epub 2020 May 4. PMID 32380253
- [Background] Barbieri E, Sestili P. Reactive oxygen species in skeletal muscle signaling. J Signal Transduct. 2012;2012:982794. doi: 10.1155/2012/982794. Epub 2011 Dec 5. PMID 22175016
- [Background] Sakellariou GK, Jackson MJ, Vasilaki A. Redefining the major contributors to superoxide production in contracting skeletal muscle. The role of NAD(P)H oxidases. Free Radic Res. 2014 Jan;48(1):12-29. doi: 10.3109/10715762.2013.830718. Epub 2013 Oct 7. PMID 23915064
- [Background] Powers SK, Ji LL, Kavazis AN, Jackson MJ. Reactive oxygen species: impact on skeletal muscle. Compr Physiol. 2011 Apr;1(2):941-69. doi: 10.1002/cphy.c100054. PMID 23737208
- [Background] Orsavova J, Misurcova L, Ambrozova JV, Vicha R, Mlcek J. Fatty Acids Composition of Vegetable Oils and Its Contribution to Dietary Energy Intake and Dependence of Cardiovascular Mortality on Dietary Intake of Fatty Acids. Int J Mol Sci. 2015 Jun 5;16(6):12871-90. doi: 10.3390/ijms160612871. PMID 26057750
- [Background] Liguori I, Russo G, Curcio F, Bulli G, Aran L, Della-Morte D, Gargiulo G, Testa G, Cacciatore F, Bonaduce D, Abete P. Oxidative stress, aging, and diseases. Clin Interv Aging. 2018 Apr 26;13:757-772. doi: 10.2147/CIA.S158513. eCollection 2018. PMID 29731617
- [Background] Mironczuk-Chodakowska I, Witkowska AM, Zujko ME. Endogenous non-enzymatic antioxidants in the human body. Adv Med Sci. 2018 Mar;63(1):68-78. doi: 10.1016/j.advms.2017.05.005. Epub 2017 Aug 17. PMID 28822266
- [Background] Romero AC. et al. 2013, 'The Exogenous Antioxidants', in J. A. Morales-González (ed.), oxidative Stress and Chronic Degenerative Diseases - A Role for Antioxidants, IntechOpen, London. doi: 10.5772/52490.
- [Background] Romeu M, Aranda N, Giralt M, Ribot B, Nogues MR, Arija V. Diet, iron biomarkers and oxidative stress in a representative sample of Mediterranean population. Nutr J. 2013 Jul 16;12:102. doi: 10.1186/1475-2891-12-102. PMID 23866833
- [Background] Tan BL, Norhaizan ME. Effect of High-Fat Diets on Oxidative Stress, Cellular Inflammatory Response and Cognitive Function. Nutrients. 2019 Oct 25;11(11):2579. doi: 10.3390/nu11112579. PMID 31731503
- [Background] Askari G, Ghiasvand R, Feizi A, Ghanadian SM, Karimian J. The effect of quercetin supplementation on selected markers of inflammation and oxidative stress. J Res Med Sci. 2012 Jul;17(7):637-41. PMID 23798923
- [Background] Buonocore D, Verri M, Giolitto A, Doria E, Ghitti M, Dossena M. Effect of 8-week n-3 fatty-acid supplementation on oxidative stress and inflammation in middle- and long-distance running athletes: a pilot study. J Int Soc Sports Nutr. 2020 Nov 11;17(1):55. doi: 10.1186/s12970-020-00391-4. PMID 33176827
- [Background] Mozaffarian D, Rimm EB. Fish intake, contaminants, and human health: evaluating the risks and the benefits. JAMA. 2006 Oct 18;296(15):1885-99. doi: 10.1001/jama.296.15.1885. PMID 17047219
- [Background] Misurcova L, Ambrozova J, Samek D. Seaweed lipids as nutraceuticals. Adv Food Nutr Res. 2011;64:339-55. doi: 10.1016/B978-0-12-387669-0.00027-2. PMID 22054960
- [Background] Dhavamani S, Poorna Chandra Rao Y, Lokesh BR. Total antioxidant activity of selected vegetable oils and their influence on total antioxidant values in vivo: a photochemiluminescence based analysis. Food Chem. 2014 Dec 1;164:551-5. doi: 10.1016/j.foodchem.2014.05.064. Epub 2014 May 22. PMID 24996369
- [Background] Yildirim E, Cinar M, Yalcinkaya I, Ekici H, Atmaca N, Guncum E. Effect of cocoa butter and sunflower oil supplementation on performance, immunoglobulin, and antioxidant vitamin status of rats. Biomed Res Int. 2014;2014:606575. doi: 10.1155/2014/606575. Epub 2014 Jul 16. PMID 25136602
- [Background] Petraru A, Ursachi F, Amariei S. Nutritional Characteristics Assessment of Sunflower Seeds, Oil and Cake. Perspective of Using Sunflower Oilcakes as a Functional Ingredient. Plants (Basel). 2021 Nov 17;10(11):2487. doi: 10.3390/plants10112487. PMID 34834848
- [Background] Kim JG, Yousef AE, Dave S. Application of ozone for enhancing the microbiological safety and quality of foods: a review. J Food Prot. 1999 Sep;62(9):1071-87. doi: 10.4315/0362-028x-62.9.1071. PMID 10492485
- [Background] El-Hamidi M. Zaher FA. Production of vegetable oils in the world and in Egypt: An overview. Bull Natl Res Cent. 2018, 42, 1-9. doi: 10.1186/s42269-018-0019-0.
- [Background] Ainsworth BE, Haskell WL, Herrmann SD, Meckes N, Bassett DR Jr, Tudor-Locke C, Greer JL, Vezina J, Whitt-Glover MC, Leon AS. 2011 Compendium of Physical Activities: a second update of codes and MET values. Med Sci Sports Exerc. 2011 Aug;43(8):1575-81. doi: 10.1249/MSS.0b013e31821ece12. PMID 21681120
- [Result] Reid MB. Invited Review: redox modulation of skeletal muscle contraction: what we know and what we don't. J Appl Physiol (1985). 2001 Feb;90(2):724-31. doi: 10.1152/jappl.2001.90.2.724. PMID 11160074